CLINICAL TRIAL: NCT04716465
Title: Dysautonomia in Patients Post COVID-19 Infection
Acronym: DYSCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moens Maarten (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: DYSCO
Record Dates: First submitted 2021-01-18; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 infected patients: In this study male and female patients who were previously infected with covid-19 (symptomatic and asymptomatic) will be included. Patients will only be eligible if they had a positive covid-19 test before inclusion in the study. More specifically, only patients who had a positive COVID-19 test 2 to 8 weeks before study inclusion are eligible.
  Interventions: Other: Dysautonomia

INTERVENTIONS:
Other: Dysautonomia — Indicators of dysautonomia

SUMMARY:
The aim for this study is further to elucidate the presence of dysautonomia in post-covid-19 patients, by evaluating heart rate variability.

DETAILED DESCRIPTION:
The COVID-19 pandemic is currently a serious global public health concern. This disease is caused by a novel coronavirus which was first discovered in Wuhan, China in 2019 and later spread rapidly throughout the world. Symptoms of the disease can manifest as fever, cough, encephalitis, myalgia, fatigue, muscle weakness, arthralgia, anosmia, and impairment in other bodily functions in the acute phase. In 17% to 67% of cases, COVID-19 patients will develop acute respiratory distress syndrome (ARDS) and critical illness. Besides the impact on the respiratory system, coronaviruses have an effect on other systems including the central nervous system, cardiovascular system, musculoskeletal system, and gastrointestinal system.

Potential long-term secondary effects on the musculoskeletal system such as muscle weakness, decreased muscle mass, and myopathies have been brought under attention. Persisting symptoms in patients recovered from COVID-19 infection are frequently a complaint with at least 1 symptom, particularly fatigue and dyspnea. In recent papers, the authors commented on the potential role of dysautonomia in the post-covid-19 entity related to microangiopathy and endothelial injury. Such lesions were already reported in brain biopsy samples of severe COVID-19.

Therefore, the aim of this study is further to elucidate the presence of dysautonomia in post-covid-19 patients, by evaluating heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosed covid-19 infection that took place 2-8 weeks before study inclusion.
* Cognitive and language functioning enabling coherent communication between the researcher and the participant.
* French-or Dutch speaking persons.

Exclusion Criteria:

* Covid-19 infection > 8 weeks ago.
* The presence of one or more coexisting conditions known to affect HRV analysis (including but not limited to atrial fibrillation, numerous atrial or ventricular extra beats, paced rhythm, left ventricular bundle branch block, cancer, kidney or hepatic failure, and diabetes mellitus)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients who were previously infected with covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  Heart rate variability will be measured using a 2-lead ECG.

SECONDARY OUTCOMES:
Electrodermal activity | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  Electrodermal activity will be measured by applying two skin conductance sensors.
Respiration rate | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  Respiration will be measured using a respiration sensor (an elastic belt) .
Blood volume pulse | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  The blood volume pulse sensor uses fingertip photo plethysmography.
Functionality and disability | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  Functional status will be evaluated by the Post-COVID-19 Functional Status Scale.
Functionality and disability | The change between baseline, 3 months (primary time endpoint), 6 months and 12 months
  Level of dyspnea during activities of daily living will be evaluated by the London chest Activity of Daily Living scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium